CLINICAL TRIAL: NCT00624104
Title: VLDL-triglyceride Under Acute Hyperinsulinaemia
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: ES-0001
Record Dates: First submitted 2008-02-18; First posted 2008-02-26 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2011-11

CONDITIONS: Obesity
Keywords: VLDL; Kinetics; Hyperinsulinaemia; Obesity
MeSH Terms: conditions — Obesity; Hyperinsulinism | interventions — Food

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — specimen of muscle specimen of adipose tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Lean male
  Interventions: Dietary Supplement: Food (fat free meal)
- 2: Males with type 2 diabetes
  Interventions: Dietary Supplement: Food (fat free meal)

INTERVENTIONS:
Dietary Supplement: Food (fat free meal) — Fat free meal (40% of REE)

SUMMARY:
The purpose of the study is to investigate and compare the lipid metabolism in lean and obese individuals. We want to investigate the effect of postprandial hyperinsulinaemia on VLDL-triglyceride metabolism

ELIGIBILITY:
Inclusion Criteria:

- Written consent

Exclusion Criteria:

* Known diseases
* Alcohol abuse
* Smoker
* Regular use of medicine

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Males with diabetes from departments out-patient clinic. Control group of healthyt volunteers
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2008-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
VLDL metabolism | Few hours

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endocrinology M, Aarhus Hospital, Aarhus C, Denmark